CLINICAL TRIAL: NCT01470859
Title: a Pilot Follow-up Study of Investigating the Effect of Pramipexole on Metabolic Network Activity Compared With Levodopa in Chinese Patients With Early Parkinson's Disease
Brief Title: The Effect of Pramipexole on Metabolic Network Activity Compared With Levodopa in Early Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Jian Wang, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2011-283
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: De Novo parkinson's disease; initial treatment; pramipexole; Levodopa; Parkinson's disease-related spatial covariance pattern
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole; carbidopa, levodopa drug combination; Levodopa; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pramipexole (Active Comparator): 0.375mg-4.5mg/day, flexible dosage according to an optimal improvement of movement dysfunction in PD patients
  Interventions: Drug: pramipexole
- Levodopa (Active Comparator): Sinemet CR CR， Controlled Release
  Interventions: Drug: Sinemet CR

INTERVENTIONS:
Drug: pramipexole — tablets, 0.375mg-4.5mg/day divided by 3 times according to the optimal improvement of motor dysfunction in PD patients. duration is 1 year.
  Other Names: Sifrol
  Arms: pramipexole
Drug: Sinemet CR — tablet of Sinemet CR, dosage of levodopa ranging from 200mg-600mg/day divided by 2 or 3 times, Duration is 1 year
  Other Names: Sinemet CR 250' (Levodopa 200mg, and 50mg carbidopa)
  Arms: Levodopa

SUMMARY:
Levodopa and non-ergot dopaminergic agonists such as pramipexole are both recommended as the first-line symptomatic treatment for early untreated Parkinson's disease (PD), previous clinical trial indicated that initial pramipexole owns advantage over levodopa regarding motor complications, on the contrary, less adverse effect like freezing and severe somnolence favors initial treatment of levodopa. Thus, it remains controversial that initiation of which medication will be better for those patients with early PD.

Parkinson's disease-related spatial covariance patter (PDRP) is a new biomarker which can represent the network activity of brain and severity of PD. Based on the literatures and our previous data, the investigators hypothesize that PDRP will be served as a biomarker to help us evaluate and compare the effect of levodopa or pramipexole on the progression of PD, which might be able to provide further evidence for clinicians to address the above critical issue.

DETAILED DESCRIPTION:
CALM-PD study found that Pramipexole can reduce the occurrence of motor complication compared with Levodopa used as initiative treatment, but it still remains debatable that initiation of which medication will be better for those patients with De Novo PD.

PDRP (Parkinson's disease-related spatial covariance pattern) is a biomarker which can represent the network activity of cortico-striato-pallido-thalamocortical pathways and highly reproducible with stable network activity in individual subjects. The study published in "J Neuroscience" in 2010 showed that the abnormal PDRP antecede the appearance of motor signs by about 2 years, indicating PDRP might be a very promising biomarker for identifying PD at its early stage. Moreover, PDRP is able to represent the progression and severity of PD as well. It was reported that Levodopa can reduce the PD-related network activity, and the degree of network suppression correlates with the clinical improvement. However, there is no study currently showing the impact of pramipexole on brain PDRP network compared with levodopa as initiative treatment.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's disease meeting United Kingdom (UK) brain bank criteria
* De Novo
* Hoehn&Yahr staging (H&Y) I-II

Exclusion Criteria:

* Atypical Parkinsonism
* Pregnant or breast-feeding women
* those with abnormal Liver/kidney function
* those participating other clinical trials within 30 days before being enrolled for this trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Izumi Y, Sawada H, Yamamoto N, Kume T, Katsuki H, Shimohama S, Akaike A. Novel neuroprotective mechanisms of pramipexole, an anti-Parkinson drug, against endogenous dopamine-mediated excitotoxicity. Eur J Pharmacol. 2007 Feb 28;557(2-3):132-40. doi: 10.1016/j.ejphar.2006.11.011. Epub 2006 Nov 14. PMID 17161393
- [Background] Parkinson Study Group. A randomized placebo-controlled trial of rasagiline in levodopa-treated patients with Parkinson disease and motor fluctuations: the PRESTO study. Arch Neurol. 2005 Feb;62(2):241-8. doi: 10.1001/archneur.62.2.241. PMID 15710852
- [Background] Huang C, Tang C, Feigin A, Lesser M, Ma Y, Pourfar M, Dhawan V, Eidelberg D. Changes in network activity with the progression of Parkinson's disease. Brain. 2007 Jul;130(Pt 7):1834-46. doi: 10.1093/brain/awm086. Epub 2007 Apr 30. PMID 17470495
- [Background] Ma Y, Tang C, Spetsieris PG, Dhawan V, Eidelberg D. Abnormal metabolic network activity in Parkinson's disease: test-retest reproducibility. J Cereb Blood Flow Metab. 2007 Mar;27(3):597-605. doi: 10.1038/sj.jcbfm.9600358. Epub 2006 Jun 28. PMID 16804550
- [Background] Tang CC, Poston KL, Dhawan V, Eidelberg D. Abnormalities in metabolic network activity precede the onset of motor symptoms in Parkinson's disease. J Neurosci. 2010 Jan 20;30(3):1049-56. doi: 10.1523/JNEUROSCI.4188-09.2010. PMID 20089913
- [Background] Wang J, Ma Y, Huang Z, Sun B, Guan Y, Zuo C. Modulation of metabolic brain function by bilateral subthalamic nucleus stimulation in the treatment of Parkinson's disease. J Neurol. 2010 Jan;257(1):72-8. doi: 10.1007/s00415-009-5267-3. Epub 2009 Aug 7. PMID 19662326

RESULTS

PARTICIPANT FLOW:
Groups:
- Levodopa: Sinemet Controlled Release (CR)
  Sinemet CR: tablet of Sinemet CR, dosage of levodopa ranging from 200mg-600mg/day divided by 2 or 3 times, Duration is 1 year
Period: Overall Study
Arm/Group | Levodopa | Pramipexole
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Levodopa: Sinemet CR
  Sinemet CR: tablet of Sinemet CR, dosage of levodopa ranging from 200mg-600mg/day divided by 2 or 3 times, Duration is 1 year
- Total: Total of all reporting groups
Arm/Group | Pramipexole | Levodopa | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.87 (5.68) | 61.9 (6.66) | 62.9 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  China | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Change of Brain Network Activity
Description: The brain network activity is evaluated by Parkinson's disease-related spatial covariance pattern(PDRP) value (Z score).
  The change of brain network activity is calculated by the PDRP value (Z score) at V5 - the PDRP value (Z score) at V1.
Time Frame: twice, baseline and 1 year after baseline
Measure: Mean (Standard Deviation); unit: Z-score in PDRP
Arm/Group | Levodopa | Pramipexole
Number analyzed (Participants) | 14 | 15
Z-score in PDRP
  Change from baseline (V5-V1) | 0.41 (0.70) | 0.61 (0.68)
  Z score at baseline (V1) | 2.21 (1.54) | 3.61 (1.77)
  Z score at 1 year (V5) | 2.29 (1.24) | 4.09 (1.07)
Statistical Analysis 1: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.84, t-test, 2 sided — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent sample t-test The statistical analysis was performed on the changes of PDRP Z score between levodopa and pramipexole groups
Statistical Analysis 2: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.93, t-test, 2 sided — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent sample t-test The statistical analysis was performed to compare the PDRP Z scores between levodopa and pramipexole groups at V1
Statistical Analysis 3: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.31, t-test, 2 sided — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent sample t-test The statistical analysis was performed to compare the PDRP Z scores between levodopa and pramipexole groups at V5

2. Secondary Outcome: Unified Parkinson's Disease Rating Score (UPDRS II, III)
Description: baseline (1st visit, V1), completion of dosage titration within 10 weeks after baseline (2nd visit, V2), 1 year after baseline (final visit, V5) UPDRS II score 0-52 (13 items); UPDRS III score 0-56 (14 items); The more scores,the more severe; the two scales were evaluated separately.
Time Frame: three times: baseline, 10 weeks, 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa | Pramipexole
Number analyzed (Participants) | 14 | 15
units on a scale
  UPDRS II at baseline (V1) | 7.3 (3.5) | 7.1 (2.9)
  UPDRS II (V2) | 5.8 (3.5) | 4.9 (3.3)
  UPDRS II at 1 year (V5) | 7.4 (3.5) | 8.4 (3.0)
  UPDRS III at baseline (V1) | 18.7 (7.7) | 23.1 (10.4)
  UPDRS III (V2) | 12.7 (4.2) | 20.1 (8.9)
  UPDRS III at 1 year (V5) | 19.5 (7.0) | 24.3 (8.8)
Statistical Analysis 1: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.691, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the UPDRS II scores at V1 scores between the levodopa and pramipexole groups
Statistical Analysis 2: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.706, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the UPDRS II scores at V2 scores between the levodopa and pramipexole groups
Statistical Analysis 3: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.635, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the UPDRS II scores at V5 scores between the levodopa and pramipexole groups
Statistical Analysis 4: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.341, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the UPDRS III scores at V1 scores between the levodopa and pramipexole groups
Statistical Analysis 5: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.049, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the UPDRS III scores at V2 scores between the levodopa and pramipexole groups
Statistical Analysis 6: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.874, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the UPDRS III scores at V5 scores between the levodopa and pramipexole groups

3. Secondary Outcome: Parkinson's Disease Questionnaire (PDQ39)
Description: The PDQ39 score was assessed at baseline (1st visit, V1) and 1 year after baseline (final visit, V5).
  PDQ39 score ranges from 0-156 (0-4 each item); the more score, the more severe.
Time Frame: twice baseline and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa | Pramipexole
Number analyzed (Participants) | 14 | 15
units on a scale
  PDQ39 at baseline (V1) | 19.38 (10.94) | 20.36 (16.49)
  PDQ39 at 1 year (V5) | 20.36 (16.49) | 21.07 (12.96)
Statistical Analysis 1: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.720, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the PDQ39 scores between levodopa and pramipexole group at V1
Statistical Analysis 2: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.867, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the PDQ39 scores between levodopa and pramipexole group at V5

4. Secondary Outcome: Hoehn&Yahr (H&Y) Staging
Description: The Hoehn and Yahr scale is a commonly used scale for describing how the symptoms of Parkinson's disease progress and the disease stages. Bigger numbers indicate more symptoms and disease progression. H&Y stage range from 0-5; the greater, the more severe.
  The H&Y stages of patients were evaluated at baseline (1st visit, V1), and 1 year after baseline (final visit, V5).
Time Frame: twice baseline and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa | Pramipexole
Number analyzed (Participants) | 14 | 15
units on a scale
  H&Y at baseline（V1） | 1.35 (0.42) | 1.43 (0.51)
  H&Y at 1 year（V5） | 1.65 (0.47) | 1.82 (0.54)
Statistical Analysis 1: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.793, indenpendent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the H&Y stages between levodopa and pramipexole group at V1
Statistical Analysis 2: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.430, independent U test — "p<0.05" is indicating the threshold for statistical significance for this comparison; independent U test The statistical analysis was performed to compare the H&Y stages between levodopa and pramipexole groups at V5

5. Secondary Outcome: Patients With Clinical Improvement as Evaluated by Global Impression Scale (CGI).
Description: Patients with a score <= 2 (very much or much improved in relation to baseline) are considered as clinically improved.
  The numbers of participants with clinical improvement are reported here. The completion of dosage titration within 10 weeks after baseline (visit 2) and 1 year after baseline (final visit)
Time Frame: twice, at 10 weeks(V2) and 1 year(V5)
Measure: Number; unit: participants
Arm/Group | Levodopa | Pramipexole
Number analyzed (Participants) | 14 | 15
participants
  Patients with improvement at V2 | 6 | 4
  Patients with improvement at V5 | 2 | 4
Statistical Analysis 1: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.345, Chi-squared — "p<0.05" is indicating the threshold for statistical significance for this comparison; The statistical analysis was performed to compare the clinical improvement between levodopa and pramipexole groups at V2
Statistical Analysis 2: Comparison: Levodopa vs Pramipexole; Test type: Superiority or Other; p = 0.410, Chi-squared — "p<0.05" is indicating the threshold for statistical significance for this comparison; The statistical analysis was performed to compare the clinical improvement between levodopa and pramipexole groups at V5

ADVERSE EVENTS:
Time Frame: 1 years
Arm/Group | Levodopa | Pramipexole
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 4/14 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa (N=14) | Pramipexole (N=15)
Somnolence (Nervous system disorders) | 0 | 2
Insomnia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Courbature (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
In the further study, a larger sample size and strict enrollment of early PD patients may enhance the accuracy of clinical trial conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No